CLINICAL TRIAL: NCT03619941
Title: Effects of 7-day Continuous Montmorency Tart Cherry Juice Supplementation in Metabolic Syndrome Participants: a Pilot Study
Brief Title: Continuous Tart Cherry Juice Supplementation With Metabolic Syndrome Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Terun Desai, PhD Student, University of Hertfordshire
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LMS/PGR/UH/03319
Record Dates: First submitted 2018-07-29; First posted 2018-08-08 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Hypertension
Keywords: Montmorency Tart Cherry; Anthocyanins; Polyphenols; Metabolic Syndrome; Insulin Resistance; Hypertension; Lipid Profile; Prediabetes
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Hypertension; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Montmorency Tart Cherry Juice (Experimental)
  Interventions: Dietary Supplement: Montmorency Tart Cherry Juice

INTERVENTIONS:
Dietary Supplement: Montmorency Tart Cherry Juice — 100% natural, tart Montmorency cherry concentrate (30mL) diluted with 100mL water.
  Concentrate contains no sweeteners, preservatives, flavourings or added sugar.
  Arms: Montmorency Tart Cherry Juice
Dietary Supplement: Placebo — Placebo drink attempted to match for total energy content, macronutrient content, appearance and taste of Montmorency tart cherry juice.
  Arms: Placebo

SUMMARY:
The present study examined the effect of Montmorency tart cherry juice on functional and blood-based cardio-metabolic markers in humans with Metabolic Syndrome. Participants consumed Montmorency tart cherry juice or a placebo beverage continuously for 7 days in a randomised, crossover trial. Outcome variables were measured immediately prior to supplementation and post-supplementation. Furthermore, on the 7th day of supplementation outcome variables were measured pre- and up to 5 hours post-bolus. It was hypothesised that Montmorency tart cherry juice would improve cardio-metabolic markers, particularly fasting insulin and systolic blood pressure. Furthermore, the study aimed to identify the mechanism of action for any effects of Montmorency tart cherry juice on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Meet 3 of 5 criteria for Metabolic Syndrome based on National Cholesterol Education Program-Adult Treatment Panel III guidelines:

1. Waist Circumference: >102cm (men), >88cm (women)
2. Fasting Serum Triglycerides: ≥1.69 mmol.L-1
3. Fasting High Density Lipoprotein: <1.03 mmol.L-1 (men), <1.29 mmol.L-1 (women)
4. Blood Pressure: ≥130 mmHg SBP or ≥85 mmHg DBP
5. Fasting Plasma Glucose: ≥6.1 mmol.L-1

Exclusion Criteria:

* Smokers
* Current or previous history of gastrointestinal, cardiovascular, hepatic or renal disease
* Currently diagnosed with diabetes or uncontrolled hypertension (≥160/100 mmHg)
* Allergy to fructose, maltodextrin or specific fruit products
* Currently taking medication (such as steroids, NSAIDs, antibiotics, antihypertensive, hypoglycaemic, lipid-lowering drugs)
* Currently using any nutritional or antioxidant supplement. Heavy alcohol consumption (>14 units per week).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Insulin | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (1 hour, 3 hour, 5 hour)
Change in Systolic and Diastolic Blood Pressure | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour)
Change in Fasting Lipid Profile (Total Cholesterol, HDL, Triglycerides, LDL) | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (1 hour, 3 hour, 5 hour)
Change in Fasting Glucose | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (1 hour, 3 hour, 5 hour)

SECONDARY OUTCOMES:
Change in 24-hour Ambulatory Blood Pressure | Baseline, Post-Supplementation (7 days)
  Systolic, Diastolic and Pulse Pressure will be measured
Change in HOMA2-IR, HOMA%S and HOMA%B | Baseline, Post-Supplementation (7 days)
  Homeostatic Model Assessment of Insulin Resistance, Sensitivity and Beta-cell function
Change in Pulse Wave Analysis | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour)
Change in Cardiac Haemodynamics | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour)
  Beat-by-beat cardiac output, stroke volume, heart rate, total peripheral resistance, mean arterial pressure will be measured
Change in Resting Metabolic Rate | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour)
Change in Angiotensin Converting Enzyme Inhibition activity | Baseline, Post-Supplementation (7 days) and Acute Post-Bolus (1 hour, 3 hour, 5 hour)

CONTACTS AND LOCATIONS:
Overall Officials: Terun Desai, Principal Investigator — University of Hertfordshire
Locations (1):
- University of Hertfordshire, Hatfield, Hertfordshire, United Kingdom

REFERENCES:
- [Derived] Desai T, Roberts M, Bottoms L. Effects of short-term continuous Montmorency tart cherry juice supplementation in participants with metabolic syndrome. Eur J Nutr. 2021 Apr;60(3):1587-1603. doi: 10.1007/s00394-020-02355-5. Epub 2020 Aug 12. PMID 32789528